CLINICAL TRIAL: NCT02412774
Title: Effects of Replacing Diet Beverages With Water on Type 2 Diabetic Obese Females Attending a Weight Loss Program - a Randomized, 24 Week Clinical Trial
Brief Title: Effects of Replacing Diet Beverages With Water on Weight Loss and Plasma Glucose Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-107
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes; Overweight; Obese
Keywords: diet beverages; water; diabetes; weight loss; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Diabetes Mellitus; Weight Loss; Insulin Resistance | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet Beverages (DBs) (Experimental): Diet beverages after the main meal+ Diet
  Interventions: Behavioral: DBs at the end of the main meal + Diet
- Water (Experimental): Water after the main meal+ Diet
  Interventions: Behavioral: Water at the end of the main meal+ Diet

INTERVENTIONS:
Behavioral: DBs at the end of the main meal + Diet — Subjects are asked to have 250 ml DBs at the end of their lunch as the main meal, while they are on a multidisciplinary diet plan for 24 weeks.
  Arms: Diet Beverages (DBs)
Behavioral: Water at the end of the main meal+ Diet — Subjects are asked to have 250 ml water at the end of their lunch as the main meal, while they are on a multidisciplinary diet plan for 24 weeks.
  Arms: Water

SUMMARY:
The purpose of the present study is to evaluate the effect of replacing diet beverages with water on weight loss and biochemical indicators for insulin sensitivity and cardiometabolic risk factors of diabetic obese and overweight female adults when they are in a multidisciplinary weight loss plan.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic female patient with 6.5<H1AC<7.2.
* Monotherapy with Metformin.
* 18-45 years of age.
* Body mass index (BMI) between 27-35 kg/ m².
* Consume DBs regularly during their habitual diet.
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Unwilling to change intake of beverages during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 24 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | 24 weeks
Insulin resistance (HOMA) | 24 weeks
Lipid profiles | 24 weeks
Waist circumference | 24 weeks
BMI | 24 Weeks
HA1C | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Farshchi, MD, PhD, Study Chair — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ameneh Madjd, Dr, Principal Investigator — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ian A Macdonald, Prof., Principal Investigator — School of Life Sciences, The University of Nottingham; Moira A Taylor, PhD, Principal Investigator — School of Life Sciences, The University of Nottingham; Reza Malekzadeh, Prof., Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences; Alireza Delavari, MD, Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lohner S, Kuellenberg de Gaudry D, Toews I, Ferenci T, Meerpohl JJ. Non-nutritive sweeteners for diabetes mellitus. Cochrane Database Syst Rev. 2020 May 25;5(5):CD012885. doi: 10.1002/14651858.CD012885.pub2. PMID 32449201